CLINICAL TRIAL: NCT01076582
Title: A Multi-centre, Randomized, Double-blind, Active Control, Parallel-group, 2-arm Study to Investigate the Effect of Ethinylestradiol / Drospirenone (0.02 mg/3 mg) Oral Contraception in a 24/4 Regimen Compared to Ethinylestradiol / Desogestrel (0.02 mg/0.15 mg) Oral Contraception in a 21/7 Regimen on Hormone Withdrawal Associated Symptoms in Otherwise Healthy Women After 4 Cycles of Treatment
Brief Title: Comparative Trial in Hormone Withdrawal Associated Symptoms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14567; 2009-014911-11 (EudraCT Number)
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Oral Contraceptive
Keywords: hormone withdrawal associated symptoms
MeSH Terms: interventions — drospirenone and ethinyl estradiol combination; Ethinyl Estradiol; Desogestrel; ethinyl estradiol-desogestrel combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: EE20/DRSP (YAZ, BAY86-5300)
- Arm 2 (Active Comparator)
  Interventions: Drug: Ethinylestradiol (EE) and desogestrel (DSG) (Mercilon)

INTERVENTIONS:
Drug: EE20/DRSP (YAZ, BAY86-5300) — 4 cycles of treatment / per cycle: 1 tablet (EE 0.02 mg / DRSP 3 mg) daily for 24 days followed by 1 placebo tablet daily for 4 days
  Arms: Arm 1
Drug: Ethinylestradiol (EE) and desogestrel (DSG) (Mercilon) — 4 cycles of treatment / per cycle: 1 tablet (EE 0.02 mg / DSG 0.15 mg) daily for 21 days followed by 1 placebo tablet daily for 7 days
  Arms: Arm 2

SUMMARY:
This clinical research study will examine whether an oral contraceptive pill taken with a monthly hormone-free interval of 4 days reduces hormone withdrawal associated symptoms compared to an oral contraceptive pill taken with a monthly hormone-free interval of 7 days after 4 cycles of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 18 and 35 years (inclusive)
* Smokers with a maximum age of 30 years at time of informed consent
* Healthy female subjects requesting contraception and currently using a low-dose EE containing oral contraceptives (OC) in a 21-day regimen (for at least three months) and suffering from at least two of the hormone withdrawal associated symptoms headache, pelvic pain and bloating during all three months prior the planned baseline cycle and requiring further OC use
* To be valid for randomization, the total 7-day composite score of hormone-withdrawal symptoms during the baseline cycle must show an increase of at least 50% during Day 22 - 28 versus the 21-day composite score during Day 1 - 21 (21-day score divided by three [for normalization])
* History of regular cyclic menstrual periods

Exclusion Criteria:

* Presence or a history of venous or arterial thrombotic/thromboembolic events (e.g. deep venous thrombosis, pulmonary embolism, myocardial infarction) or of a cerebrovascular accident, or presence or history of prodrome of a thrombosis (e.g. transient ischemic attack, angina pectoris) and conditions that could increase the risk to suffer from any of the above mentioned disorders, e.g., a family history indicating a hereditary predisposition. Hereditary or acquired predisposition for venous or arterial thrombosis, such as APCresistance, antithrombin-III-deficiency, protein C deficiency, protein S deficiency, hyperhomocysteinemia and antiphospholipid-antibodies (anticardiolipin-antibodies, lupus anticoagulant).
* History of migraine with focal neurological symptoms.
* Diabetes mellitus with vascular involvement.
* Obesity (Body Mass Index >32.0 kg/m2)
* Moderate to severe hypertension (repeated measurements of systolic blood pressure >140 mmHg and/or diastolic blood pressure >90 mmHg).
* Pancreatitis or a history thereof if associated with severe hypertriglyceridemia.
* Presence or history of severe hepatic disease as long as liver function values have not returned to normal.
* Jaundice and / or pruritus related to cholestasis (Gilbert´s syndrome excepted), or history of cholestatic jaundice associated with pregnancy or previous combined OC use
* Severe renal insufficiency or acute renal failure.
* Presence or history of liver tumors (benign or malignant), or known or suspected sex-steroid influenced malignancies or premalignant disease (e.g. of the genital organs or the breasts).

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 592 (Actual)
Dates: Start 2010-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline to cycle 4 in the sum of composite score during cycle days 22 - 28. The composite score comprises headache, pelvic pain and bloating (each measured by 7-point Likert scales). | Cycle days 22 - 28 of baseline cycle and cycle 4.

SECONDARY OUTCOMES:
change from baseline to cycle 4 in the sum of individual scores during cycle days 22 - 28 (AUC of days 22 - 28 for each score), | Cycle days 22 - 28 of baseline cycle and cycle 4
change from baseline to cycle 4 in number of days, where individual hormone withdrawal symptoms are present on cycle days 22 - 28 (i.e. Likert Scale >= 1), | Cycle days 22 - 28 of baseline cycle and cycle 4
change from baseline to cycle 4 in maximum intensity of individual hormone withdrawal symptoms on cycle days 22 - 28, | Cycle days 22 - 28 of baseline cycle and cycle 4
rescue medication consumption | baseline cycle and cycle 4
bleeding pattern | reference period is 90 days.
evaluation of questionnaires: Q-LES-Q (short version) | baseline cycle and cycle 4
Adverse Event collection | up to 10 days after end of cycle 4
heart rate | up to 10 days after end of cycle 4
blood pressure | up to 10 days after end of cycle 4

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (38):
- Argentina (2):
  - Buenos Aires, Ciudad Auton. de Buenos Aires
  - Rosario, Santa Fe Province
- Chile (3):
  - Santiago, Santiago Metropolitan
  - Santiago
  - Temuco
- Colombia (3):
  - Bucaramanga, Santander Department
  - Bogotá
  - Medellín
- Czechia (3):
  - Brno
  - Prague
  - Tábor
- Germany (6):
  - Heidelberg, Baden-Wurttemberg
  - Fürth, Bavaria
  - Hanover, Lower Saxony
  - Leipzig, Saxony
  - Magdeburg, Saxony-Anhalt
  - Jena, Thuringia
- Italy (3):
  - Florence
  - Milan
  - Siena
- Philippines (2):
  - Manila
  - Pasig
- Portugal (3):
  - Lisbon, Lisbon District
  - Coimbra
  - Porto
- Moscow, Russia
- South Korea (2):
  - Seoul, Korea
  - Seoul
- Switzerland (3):
  - Basel, Canton of Basel-City
  - Bern, Canton of Bern
  - Sankt Gallen, Canton of St. Gallen
- Thailand (3):
  - Bangkok, Thailand
  - Songkhla, Thailand
  - Bangkok
- United Kingdom (3):
  - Leeds, West Yorkshire
  - Liverpool
  - London
- Caracas, Venezuela

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/